CLINICAL TRIAL: NCT00002040
Title: Open, Non-Comparative Study of Intravenous and Oral Fluconazole in the Treatment of Acute Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 012L; 056-164A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Injections, Intravenous; Cryptococcosis; Fluconazole; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To evaluate the safety and effectiveness of fluconazole as an intravenous dose as initial treatment for acute cryptococcal meningitis followed by oral therapy in AIDS and non-AIDS patients. Both newly diagnosed and relapsed patients are eligible. The effectiveness of maintenance fluconazole therapy in sustaining a clinical cure in AIDS patients will also be evaluated.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antivirals such as zidovudine. Prophylaxis for Pneumocystis carinii pneumonia. Aerosolized pentamidine.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Written informed consent must be obtained for each patient, either from the patient himself or from the patient's legal guardian.

* Patient's treatment status must be one of the following:
* No prior systemic antifungal therapy for cryptococcosis.
* Relapse after prior therapy. The success of prior therapy must have been documented by negative CSF culture at the end of therapy. Following prior therapy, such patients may not have received more than 1 mg/kg/wk amphotericin B in the 4 weeks before entry into the study.

Prior Medication:

Allowed:

* Antivirals such as zidovudine (AZT). Prophylaxis for Pneumocystis carinii pneumonia. Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* A history of allergy to or intolerance of imidazoles or azoles.
* Moderate or severe liver disease defined by specified lab values.
* Life expectancy of < 2 weeks.

Concurrent Medication:

Excluded:

* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications except aerosolized pentamidine.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* A history of allergy to or intolerance of imidazoles or azoles.
* Moderate or severe liver disease defined by specified lab values.
* Life expectancy of < 2 weeks.

Prior Medication:

Excluded:

* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications except aerosolized pentamidine.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Cook County Hosp, Chicago, Illinois
  - SUNY / Health Sciences Ctr at Brooklyn, Brooklyn, New York
  - Cornell Univ Med Ctr, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania